CLINICAL TRIAL: NCT06818838
Title: A Multicenter, Open, Single-arm, Single-dose, Dose-escalation, and Expanded Phase I/II Study Evaluating the Safety, Tolerability, and Efficacy of LY-M001 Injection in Adult Patients With Type I Gaucher Disease
Brief Title: A Clinical Study Evaluating LY-M001 Injection in the Treatment of Adult Patients With Type I Gaucher Disease
Acronym: GD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lingyi Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY-M001-GD-101
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gaucher Disease Type 1
Keywords: anaemia; Gene therapy
MeSH Terms: conditions — Gaucher Disease; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I: LY-M001 Backdose (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of LY-M001 at backdose.
  Interventions: Genetic: LY-M001
- Phase I: LY-M001 Dose group 1 (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of LY-M001 at dose group 1.
  Interventions: Genetic: LY-M001
- Phase I: LY-M001 Dose group 2 (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of LY-M001 at dose group 2.
  Interventions: Genetic: LY-M001
- Phase II: LY-M001 at the recommended dose (Experimental): Participants receive a single, peripheral IV infusion of LY-M001 at the recommended dose.
  Interventions: Genetic: LY-M001

INTERVENTIONS:
Genetic: LY-M001 — Single Intravenous Infusion of LY-M001 Injection.

SUMMARY:
Gaucher disease (GD) is caused by mutations in the GBA1 gene, which leads to a lack or reduction of GCase activity. The consequences of this deficiency are generally attributed to the accumulation of the GCase substrate, Glucosylceramide (GlcCer), in macrophages in the liver, spleen, kidney, bone, lung, and even the brain, inducing their transformation into Gaucher cells whose cell cytoplasm presenting a characteristic "crumpled tissue paper" appearance, leading to pathological changes in involved tissues and organs.LY-M001 Injection is an rAAV8 vector gene therapy product. It can specifically transduce the target organ liver after a single intravenous administration and express the GCase protein in liver cells for a long period of time.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, efficacy, immunogenicity, pharmacokinetics and pharmacokinetics of LY-M001 injection in patients with GD1 using a multicenter, open, single-arm, single-dose, dose-escalation and extended clinical design. This study includes the main study phase and the long-term follow-up study phase. The primary study period is 52 weeks after LY-M001 infusion, and the long-term follow-up period is 53 weeks to 5 years after LY-M001 infusion.Subjects who complete the 52 weeks follow up period or who prematurely withdraw in this study will enter the long-term follow-up study phase to obtain long-term assessment data.

Phase I is a dose escalation study consists of three preset dose groups, including one rollback dose group and two incremental dose groups, which are: Backdose (5 × 10^12 vg/kg) group, dose group 1 (1.5 × 10^13 vg/kg) and dose group 2 (3.0 × 10^13 vg/kg), where dose group 1 was the starting dose of the Phase I study. Three subjects are enrolled in each dose group one by one, and each subject is added to the next subject after at least 28 days of DLT observation to determine safety. Phase I studies enrolled approximately 6 to 12 (up to 12) evaluable subjects.

Phase II is a dose expansion study. After all subjects in Phase I study have completed the Day 28 (D28) observation following LY-M001 infusion, the Recommended Phase 2 Dose (RP2D) will be determined by the Safety Review Committee (SRC), which will also decide whether to proceed to the dose-expansion Phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 60 years, male or female.
2. The subjects should fully understand the purpose, nature, and method of this study as well as possible adverse reactions, and sign the informed consent form (ICF) voluntarily.
3. Patients with confirmed double mutations in the GBA1 allele through laboratory testing, and the glucocerebrosidase activity was reduced to less than 30% of the normal value(For example, the result of the dried blood spot (DBS) method is < 1.19 μmol/L/h), and meeting the standard clinical diagnosis criteria for GD1.
4. Patients who meet a) or b) below:

   1. Treated patients with Gaucher disease type I who had previously received enzyme replacement therapy (ERT) or substrate clearance therapy (SRT) with GD, were on stable medication, eluted 5 drugs for a half-life or more before administration, or were comprehensively judged to be stable by the investigator.
   2. Newly treated or untreated GD1 patients who meet one or more of the following criteria at screening:

      * Hemoglobin ≥80g/L and less than the lower limit of normal;
      * Platelets ≥40×10^9/L and less than the lower limit of normal;
      * Hepatomegaly;
      * Splenomegaly.
5. Negative pregnancy test for female subjects of childbearing potential (WOCBP). Notes: WOCBP is defined as the absence of postmenopausal status (continuous amenorrhea of at least 12 months with no identifiable cause other than menopause), and the absence of surgical (i.e., ovarian, salpingectomy, and/or hysterectomy) or Investigator-determined cause of permanent infertility due to other causes (e.g., lenticular hypoplasia) after menarche in female subjects.
6. Subjects and their partners have no childbearing plans from the screening period to 6 months after the end of the study, and voluntarily adopt effective contraceptive measures (e.g., abstinence, condoms, etc.); subjects have no plans to donate sperm or eggs.
7. Subjects are not to donate blood during the study and for at least 1 year after the end of the study.

Exclusion Criteria:

1. AAV8 neutralizing antibody positive (Antibody titer > 1:40).
2. Patients with clinically diagnosed Gaucher disease type II or III (GD2 or GD3).
3. Active and progressive bone disease that is expected to require surgical treatment within the next 6 months.
4. Subject has idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), thrombocytopenia, anemia, hepatomegaly, splenomegaly, and/or osteoporosis unrelated to GD as judged by the Investigator.
5. Treatment or disposal of investigational drugs or investigational devices received in other clinical studies within 28 days prior to screening or within 5 half-lives (drugs only), whichever is older.
6. Evidence of clinically significant liver disease, fragile liver, or history of exposure to hepatotoxins that meets, but is not limited to, any of the following at the time of screening:

   * Progressive hepatomegaly larger than 3 times the normal volume.
   * History of stage 2 or above liver fibrosis.
   * AST, ALT, or TBIL are 1.5 times higher than ULN.
   * A history of alcohol or drug abuse within the previous 2 years (defined as having consumed more than 14 standard units of alcohol per week [1 standard unit containing 14 g of alcohol, such as 360 mL beer, 45 mL spirits containing 40% or more alcohol, or 150 mL wine]).
   * Hepatitis B surface antigen (HBsAg) positive and HBV deoxyribonucleic acid (HBV-DNA) positive (HBV-DNA>10^3 copy number /mL); Or take hepatitis B drugs (such as interferon, lamivudine, adefovir and entecavir); Or antibodies to hepatitis C virus (HCV) and positive for hepatitis C virus RNA.
7. Human immunodeficiency virus (HIV) antibody positive or Treponema pallidum antibody positive.
8. Severe hyperlipidemia (triglycerides > 11.29mol/L).
9. Uncontrolled concomitant or infectious diseases (need to be determined by the investigator based on clinical practice).
10. The subject has received or plans to receive bone marrow transplantation, hematopoietic stem cell transplantation and/or major organ transplantation, including but not limited to liver transplantation, kidney transplantation, etc.
11. Subject has received erythropoietin, transfusion, or red blood cell transfusion within 3 months prior to screening; or platelet transfusion within 1 month prior to screening.
12. Clinically diagnosed or investigator-determined serious cardiovascular disease (such as heart failure ≥3 from the New York College of Cardiology [NYHA]).
13. Hypersensitivity to any component of LY-M001 injection.
14. Previous treatment with any type of gene therapy or cell therapy.
15. Use of systemic immunosuppressive agents or steroid therapy other than those required by the protocol for prophylactic administration within 3 months prior to dosing.
16. History of cancer within 5 years prior to screening, or currently active neoplastic disease, except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated.
17. Has received a live attenuated vaccine within 4 months prior to screening or plans to receive a live attenuated vaccine during the clinical trial.
18. Other conditions that, in the opinion of the Investigator, make the subject unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of adverse events (AE) and serious adverse events (SAE) within 52 weeks after LY-M001 infusion | From enrollment to 52 weeks after administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Phase I: Incidence rate of dose-limiting toxicity (DLT) events determined by the data safety review committee (SRC) within at least 28 days after LY-M001 infusion. | From enrollment to 52 weeks after administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.The adverse events defined as dose-limiting toxicity (DLT) have been clearly specified in the protocol.
Phase I: Liver function levels (including alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin [TBIL], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT]) within 52 weeks after LY-M001 infusion. | From enrollment to 52 weeks after administration
  Incidence rate of liver function-related adverse events evaluated by CTCAE V5.0.
Phase II: Blood glucocerebrosidase (GCase) activity level. | From enrollment to 52 weeks after administration
  Evaluation based on the detected values of blood glucocerebrosidase（GCase).
Phase II: The incidence rates of adverse events (AEs) and serious adverse events (SAEs), as well as the occurrence of abnormalities in 12-lead electrocardiogram (ECG) findings, vital signs, laboratory test parameters, and physical examination results. | From enrollment to 52 weeks after administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Phase I: Liver volume and spleen volume (if applicable) | From enrollment to 52 weeks after administration
  1. Change from baseline in liver volume as measured by MRI through 52 weeks after infusion of LY-M001;
  2. Change from baseline in spleen volume as measured by MRI through 52 weeks after infusion of LY-M001.
Phase I: Hemoglobin levels | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in hemoglobin levels through 52 weeks after infusion of LY-M001.
Phase I:Bone mineral density (BMD) after administration | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in bone mineral density (BMD) by dual-energy X-ray absorptiometry through 52 weeks after infusion of LY-M001.
Phase I: Glucocerebrosidase (GCase) protein levels in blood | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in GCase protein levels through 52 weeks after infusion of LY-M001.
Phase I: Glucosylsphingosine (Lyso-GL1) in blood | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in Lyso-GL1 levels in blood through 52 weeks after infusion of LY-M001.
Phase I: Platelet count | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in platelet count through 52 weeks after infusion of LY-M001.
Phase I: Bone marrow burden (BMB) after administration | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in bone marrow burden as measured by MRI through 52 weeks after infusion of LY-M001.
Phase I: Glucocerebrosidase (GCase) enzyme activity levels in blood | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in GCase enzyme activity levels in blood through 52 weeks after infusion of LY-M001.
Phase II: Glucocerebrosidase (GCase) protein levels in blood | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in GCase protein levels in blood through 52 weeks after infusion of LY-M001.
Phase II: Glucosylsphingosine (Lyso-GL1) in blood | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in Lyso-GL1 levels in blood through 52 weeks after infusion of LY-M001.
Phase II: Liver volume and spleen volume (if applicable) | From enrollment to 52 weeks after administration
  1. Change from baseline in liver volume as measured by MRI through 52 weeks after infusion of LY-M001;
  2. Change from baseline in spleen volume as measured by MRI through 52 weeks after infusion of LY-M001.
Phase II: Hemoglobin levels | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in hemoglobin levels through 52 weeks after infusion of LY-M001.
Phase II: Platelet count | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in platelet count through 52 weeks after infusion of LY-M001.
Phase II: Bone mineral density (BMD) | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in bone mineral density by dual-energy X-ray absorptiometry through 52 weeks after infusion of LY-M001.
Phase II: Bone marrow burden (BMB) | From enrollment to 52 weeks after administration
  Evaluate the change from baseline in bone marrow burden as measured by MRI through 52 weeks after infusion of LY-M001.

CONTACTS AND LOCATIONS:
Overall Officials: Fengkui Zhang, PhD, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
The study is in its early stages and will consider releasing data and related information when detailed and sufficient safety and efficacy data are available in subjects.